CLINICAL TRIAL: NCT04198129
Title: The Evaluation of Postoperative Antibiotics in Non-Infected Mandible Fractures
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nagi Demian, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0640
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-02

CONDITIONS: Jaw Fractures; Infection
Keywords: Infection; Jaw fracture
MeSH Terms: conditions — Jaw Fractures; Infections | interventions — sultamicillin; Clindamycin; Amoxicillin-Potassium Clavulanate Combination; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Trial groups will receive a single post-operative dose administration of Unasyn 3g or Clindamycin 600mg (for penicillin allergies), then the patients in the trial group will be switched to oral Augmentin 875mg twice a day for 7 days (Amoxicillin and Clavulanic acid which is clinically interchangeable with Unasyn), or oral Clindamycin 150mg to 300mg four times a day for 7 days (for penicillin allergies). If the patient is discharged home prior to completing 7 days of oral antibiotic therapy, patient will receive prescription to finish the remaining doses of antibiotics for a total period of 7 days.
  Interventions: Drug: Antibiotic treatment (Unasyn or Cleocin); Drug: Antibiotic treatment (Augmentin or Cleocin)
- Control (Active Comparator): Control group will not receive any postoperative antibiotics other than what is accepted as preoperative prophylactic antibiotics as per current standards of care.
  Interventions: Other: Control Group

INTERVENTIONS:
Drug: Antibiotic treatment (Unasyn or Cleocin) — Trial groups will receive a single post-operative dose administration of Unasyn 3g or Clindamycin 600mg (for penicillin allergies)
  Other Names: UNasyn is the trade name and the genric name is Ampicillin and Sub lactam. Cleocin is a trade name and the generic name is clindamycin.
  Arms: Treatment
Drug: Antibiotic treatment (Augmentin or Cleocin) — the patients in the trial group will be switched to oral Augmentin 875mg twice a day for 7 days, or oral Clindamycin 150mg to 300mg four times a day for 7 days (for penicillin allergies).
  Other Names: Augmentin is the trade name and the generic is Amoxicillin Clavulinate or clavulinic acid. Cleocin is the trade name and the generic is clindamycin.
  Arms: Treatment
Other: Control Group — Control group will not receive any postoperative antibiotics other than what is accepted as preoperative prophylactic antibiotics as per current standards of care
  Arms: Control

SUMMARY:
The purpose of the study is to evaluate if postoperative antibiotic use in patients with mandible trauma reduce the risk of postoperative infections and does the benefit differ based on severity, soft tissue loss, other concomitant injuries, and medical problems

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of antibiotics postoperatively in non-infected mandible fractures compared to the lack of postoperative antibiotics in the same population.

The first outcome measure is infection. Evidence of infection includes persistent swelling, fever, recurrent swelling, erythema, and purulent discharge.

The second outcome measure is no infection. Absence of persistent swelling, fever, recurrent swelling, erythema, and purulent discharge.

Outcome measures will be assessed on follow-up visits: post op week 1, post op week 3, and post op week 6-8. Latest follow-up is up to 8 weeks. If the subject presents with any of the above mentioned symptoms during the 8 week post-op period, the subject will be considered positive for infection.

Prospective randomized trial: Control group will not receive any postoperative antibiotics other than what is accepted as preoperative prophylactic antibiotics as per current standards of care. Trial groups will receive a single post-operative dose administration of Unasyn 3g or Clindamycin 600mg (for penicillin allergies), then the patients in the trial group will be switched to oral Augmentin 875mg twice a day for 7 days (Amoxicillin and Clavulanic acid which is clinically interchangeable with Unasyn), or oral Clindamycin 150mg to 300mg four times a day for 7 days (for penicillin allergies). If the patient is discharged home prior to completing 7 days of oral antibiotic therapy, patient will receive prescription to finish the remaining doses of antibiotics for a total period of 7 days.

The patient will follow up post op week 1, post op week 3, and post op week 6-8. Latest follow-up is up to 8 weeks.

Patients will be monitored for any complications, including reaction to IV and oral antibiotics. Patient will assessed after the one-time post-op IV antibiotic dose and during their follow-up visits at weeks 1, 3, and 6-8.

ELIGIBILITY:
Inclusion Criteria:

* All mandible fracture patients planned for Open Reduction and Internal Fixation (ORIF)

Exclusion Criteria:

* Age - < 18 years
* Pregnancy
* Fracture Site - closed / non-dentate eg. Condylar neck, edentulous
* Soft Tissue Injury - > Grade 4 (GSW)
* Allergic to all study drugs
* Medical Problems

  1. Diabetes - Hb A1C > 10
  2. Immunologic compromise
  3. On Chemotherapy
* Interval - Injury to Surgery - > 10days
* Already receiving antibiotics for

  1. Another wound eg. Open fracture prophylaxis
  2. Documented / suspected infection
* Inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Evidence of infection as measured by presence of persistent swelling, | post treatment week1
Evidence of infection as measured by presence of persistent swelling, | post treatment week 3
Evidence of infection as measured by presence of persistent swelling, | post treatment week 6-8
Evidence of infection as measured by presence of fever | post treatment week 1
Evidence of infection as measured by presence of fever | post treatment week 3
Evidence of infection as measured by presence of fever | post treatment week 6-8
Evidence of infection as measured by presence of recurrent swelling | post treatment week 1
Evidence of infection as measured by presence of recurrent swelling | post treatment week 3
Evidence of infection as measured by presence of recurrent swelling | post treatment week 6-8
Evidence of infection as measured by presence of erythema | post treatment week 1
Evidence of infection as measured by presence of erythema | post treatment week 3
Evidence of infection as measured by presence of erythema | post treatment week 6-8
Evidence of infection as measured by presence of purulent discharge | post treatment week 1
Evidence of infection as measured by presence of purulent discharge | post treatment week 3
Evidence of infection as measured by presence of purulent discharge | post treatment week 6-8

SECONDARY OUTCOMES:
No evidence of infection as measured by absence of persistent swelling | post treatment week 1
No evidence of infection as measured by absence of persistent swelling | post treatment week 3
No evidence of infection as measured by absence of persistent swelling | post treatment week 6-8
No evidence of infection as measured by absence of fever | post treatment week 1
No evidence of infection as measured by absence of fever | post treatment week 3
No evidence of infection as measured by absence of fever | post treatment week 6-8
No evidence of infection as measured by absence of recurrent swelling | post treatment week 1
No evidence of infection as measured by absence of recurrent swelling | post treatment week 3
No evidence of infection as measured by absence of recurrent swelling | post treatment week 6-8
No evidence of infection as measured by absence of erythema | post treatment week 1
No evidence of infection as measured by absence of erythema | post treatment week 3
No evidence of infection as measured by absence of erythema | post treatment week 6-8
No evidence of infection as measured by absence of purulent discharge | post treatment week 1
No evidence of infection as measured by absence of purulent discharge | post treatment week 3
No evidence of infection as measured by absence of purulent discharge | post treatment week 6-8

CONTACTS AND LOCATIONS:
Overall Officials: Nagi Demian, DDS/MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - Memorial Hermann Hospital, Houston, Texas
  - Th University of Texas Health Science Center at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No